CLINICAL TRIAL: NCT05336422
Title: Sun Exposure of Outdoor Workers in Mayotte and Reunion Island
Acronym: EXTRASOL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021/CHU/38
Record Dates: First submitted 2022-03-14; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Sun Exposure
Keywords: workers; sun exposure
MeSH Terms: interventions — Radiometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- training on the risks associated with sun exposure (Experimental): power point on the risks associated with sun exposure
  Interventions: Other: training on the risks associated with sun exposure

INTERVENTIONS:
Other: training on the risks associated with sun exposure — 15-minute power point and presentation on the risks of sun exposure
  Other Names: dosimetry

SUMMARY:
The UV index in Mayotte and Reunion is greater than 14, eight months out of twelve. This index decreases linearly over the period from mid-April to mid-August where it can drop to reach an index of 8 in July. The inhabitants are therefore exposed to a maximum intensity of UV radiation according to the World Health Organization (WHO).

The WHO recommends extreme precautions for indices greater than 11 (avoid exposure between 11 a.m. and 3 p.m. (GMT+3 hours), stay in the shade, wear a t-shirt, sunglasses, hat and sunscreen).

Sun exposure is a major risk factor in the development of skin cancer, basal cell cancer, squamous cell cancer and cutaneous melanoma. It is also the cause of premature aging of the skin. Furthermore, it causes ocular complications such as the occurrence of cataracts and this without distinction of skin phenotype.

There is currently no prevention campaign on the risks of sun exposure in Mayotte or Reunion for adults, while many risky behaviors are observed both in the professional field and during leisure activities. In order to better understand risk-taking and choose appropriate awareness-raising tools, it is necessary to identify the knowledge, attitudes and practices (KAP) of these populations in terms of risk of sun exposure and to measure the impact of solar prevention education actions.

ELIGIBILITY:
Inclusion Criteria:

* Live in Mayotte or Reunion island
* > 18 years old
* Work outdoors > 2 hours a day in one of the identified professions
* Belong to the list of targeted companies

Exclusion Criteria:

* Person deprived of liberty by judicial or administrative decision, minor, and person subject to a legal protection measure: guardianship or curators
* Person not agreeing to participate
* No one speaking any of the following languages: English / French / Shimaore / Kibushi / Creole or Comorian
* Person who cannot be followed during the 6 months of the study
* Inability to answer the questionnaire

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Assess the knowledge of photo-exposed workers on the risks associated with exposure to the sun. | 6 month
  knowledge quiz

SECONDARY OUTCOMES:
Assess the change in attitudes and practices of photo-exposed workers | 6 month
  attitudes and practices of photo-exposed workers quiz
fitzpatrick scale : classification of skin types (phototype I to VI) | 6 month
  phototype and knowledge level
knowledge questionnaire | 6 month
  phototype and knowledge level
Obtain UV dosimetry data by occupation to confirm risk exposure during working hours. | 6 month
  dosimetry data

CONTACTS AND LOCATIONS:
Locations (2):
- Mayotte, Chirongui, Mayotte
- Reunion, Saint-Pierre, Reunion

IPD SHARING:
Plan to Share IPD: No